CLINICAL TRIAL: NCT00086489
Title: Phase 1 Open Label, Non-Randomized, Dose Escalation Study To Evaluate The Safety, Tolerability, Pharmacokinetics, Immune Function Effects, And Efficacy Of Multiple Doses Of CP-675,206 In Patients With Advanced Melanoma, And Phase 2, Open Label, Randomized Study To Evaluate the Efficacy, Safety, Tolerability And Pharmacokinetics Of 2 Regimens Of CP-675,206 In Patients With Advanced Melanoma.
Brief Title: CP-675,206 In Patients With Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3671002
Record Dates: First submitted 2004-07-01; First posted 2004-07-05 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Malignant Melanoma
Keywords: metastatic melanoma; multiple dose
MeSH Terms: conditions — Melanoma | interventions — tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10 mg/kg (Experimental): pts treated at 10 mg/kg dose level on a monthly regimen
  Interventions: Drug: CP-675,206
- 15 mg/kg (Experimental): pts treated at 15 mg/kg dose level on a quarterly regimen
  Interventions: Drug: CP-675,206

INTERVENTIONS:
Drug: CP-675,206 — pts treated at 10 mg/kg dose level on a monthly regimen
  Arms: 10 mg/kg
Drug: CP-675,206 — pts treated at 15 mg/kg dose level on a quarterly regimen
  Arms: 15 mg/kg

SUMMARY:
The purpose of this study is to assess the efficacy, safety, and tolerability of monoclonal antibody therapy using 2 regimens for the treatment of advanced melanoma

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed: Stage III (AJCC 6th edition)xxl unresectable melanoma, with measurable disease (either locally relapsed unresectable, in-transit lesions or unresectable draining nodes) or Stage IV melanoma, including:
* Metastasis to skin, subcutaneous tissues or distant lymph nodes, or
* Metastasis to lungs, or
* Metastasis to all other visceral sites with either LDH <= ULN (upper limit of normal) or a single site of metastasis
* Note: Patients with melanoma of ocular origin will be considered ineligible
* Documented progressive disease following adjuvant therapy, localized therapy or other therapy for metastatic disease
* Measurable disease defined by at least one target lesion that can be accurately measured and whose size is at least 1.0 cm (by spiral CT) or 2.0 cm (by conventional techniques) in its longest diameter
* ECOG performance status of 0 or 1 Life expectancy of > 3 months
* Either gender, aged 18 years and above
* Adequate bone marrow, hepatic, and renal functions determined within 2 weeks prior to starting therapy, defined as:
* Absolute neutrophil count >= 1.5 x 10(9)cells/L
* Platelets >= 100 x 10(9)/L
* Hemoglobin >= 10 g/dL
* Aspartate and alanine aminotransferases (AST, ALT) <= 2.5 x ULN (<= 5 x ULN, if documented liver metastases are present)
* Total bilirubin <= 1.5 x ULN
* Creatinine <= 1.5 x ULN
* Patients must have recovered from all prior treatment related toxicities, to baseline status, or a CTC grade of 0 or 1. Post-surgical pain shall not be considered a basis for exclusion.
* Females must either be not of childbearing potential [surgically sterilized, which includes tubal ligation, or at least 2 years postmenopausal; not breastfeeding], or practicing 1 form of approved contraception for at least three months prior to entry into the study with 1 of the following methods: (a) oral contraceptives, (b) intrauterine device, (c) implanted contraceptive (such as Norplant®), (d) injected contraceptives (such as Depo-Provera®), (e) diaphragm, (f) sexual partner must use condom or be surgically sterilized, or (g) sexually inactive. Females of childbearing potential must be instructed to avoid pregnancy during study participation. Negative serum or urine pregnancy test must be documented during screening evaluation.
* Must be willing and able to provide written informed consent.

Exclusion Criteria:

* Received immunotherapy for cancer within one month prior to the start of screening
* Patients previously treated on this protocol
* History of, or significant evidence of risk for, chronic inflammatory or autoimmune disease (e.g. Addison's disease, asthma, celiac disease, multiple sclerosis, Graves Disease, Hashimoto's thyroiditis, inflammatory bowel disease, psoriasis, rheumatoid arthritis, systemic lupus erythematosus, etc.)
* Potential requirement for systemic corticosteroids or concurrent immunosuppressive drugs based on prior history.
* History of autoimmune colitis or other chronic gastrointestinal conditions associated with diarrhea or bleeding, or current acute colitis of any origin.
* Pregnant or lactating women.
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol.
* Diagnosed or suspected brain metastases. Patients with past history of brain metastases but with no radiologic evidence within 12 weeks prior to enter into the protocol will be eligible.
* Any serious uncontrolled medical disorder or active infection, which would impair their ability to receive study treatment.
* Coexisting malignancies except for basal or squamous cell carcinoma of the skin.
* Received any prior CTLA4 inhibiting agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2003-08; Primary Completion 2007-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Safety | At every scheduled visit for a maximum of 2 years from first dose of study drug
Tumor response | Assessed every 2-3 months up to 2 years from first dose of study drug

SECONDARY OUTCOMES:
Monitor for human anti-human antibodies at the end of the study | Pre-dose (Cycle 1 only) and end of study
Explore genetic influences on safety and or immune response | Pre-dose, Cycle 1
Assess PK during treatment | All cycles as pre-specified in protocol

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Research Site, Los Angeles, California
  - Research Site, Tampa, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Ann Arbor, Michigan
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas

REFERENCES:
- [Derived] Comin-Anduix B, Lee Y, Jalil J, Algazi A, de la Rocha P, Camacho LH, Bozon VA, Bulanhagui CA, Seja E, Villanueva A, Straatsma BR, Gualberto A, Economou JS, Glaspy JA, Gomez-Navarro J, Ribas A. Detailed analysis of immunologic effects of the cytotoxic T lymphocyte-associated antigen 4-blocking monoclonal antibody tremelimumab in peripheral blood of patients with melanoma. J Transl Med. 2008 May 1;6:22. doi: 10.1186/1479-5876-6-22. PMID 18452610